CLINICAL TRIAL: NCT04054297
Title: The Effect of a Low Compared to a High Glycemic Index/Saturated Fatty Acid Diet on Hepatic Fat
Brief Title: Glycemic Index/Saturated Fatty Acid Diet and Hepatic Fat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NL69685.068.19
Record Dates: First submitted 2019-08-01; First posted 2019-08-13 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Fatty Liver, Nonalcoholic; Diet, Healthy; Obesity
Keywords: NAFLD; Diet; Glycemic index
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High GI/SFA diet (Experimental): Subjects will adhere to a two-week high GI and high SFA diet. Crossover design, randomly assigned to start with either high GI/SFA or low GI/SFA. 4 week washout between the two diets.
  Interventions: Behavioral: High GI/SFA diet
- Low GI/SFA diet (Experimental): Subjects will adhere to a two-week low GI and low SFA diet. Crossover design, randomly assigned to start with either high GI/SFA or low GI/SFA. 4 week washout between the two diets.
  Interventions: Behavioral: Low GI/SFA diet

INTERVENTIONS:
Behavioral: High GI/SFA diet — Subject will adhere to a 2 week high GI/SFA diet.
  Arms: High GI/SFA diet
Behavioral: Low GI/SFA diet — Subject will adhere to a 2 week low GI/SFA diet.
  Arms: Low GI/SFA diet

SUMMARY:
Excessive fat in the liver is associated with impairments in metabolic health. Reducing the amount of carbohydrates and fat both have been shown to reduce liver fat. However, not only the amount fats and carbohydrates, but also their quality have been shown to influence liver fat. Diets high in saturated fatty acids (SFA) and diets with a high glycemic index (GI) have been shown to increase liver fat content. However, available data from human dietary intervention studies is limited and these studies did not reflect a realistic diet. In the present study a combination of low GI/SFA on the one hand and high GI/SFA on the other hand is used to reflect realistically a healthy and an unhealthy diet as they are actually consumed by the Dutch population.

The primary objective of this study is to investigate whether a two-week low compared to high GI/SFA diet reduces liver fat content. In addition, it will be investigated whether a two- week low compared to high GI/SFA diet reduces DNL, lowers the 24-hour glycemic response, lowers hepatic glycogen content, increases hepatic fat oxidation and changes hepatic lipid composition. Furthermore, the metabolic response to a meal (metabolites related to energy metabolism and substrate oxidation) will be studied upon the low and high GI/SFA diets.

DETAILED DESCRIPTION:
Rationale:

Excessive fat in the liver is associated with impairments in metabolic health. Reducing the amount of carbohydrates and fat both have been shown to reduce liver fat. However, not only the amount fats and carbohydrates, but also their quality have been shown to influence liver fat. Diets high in saturated fatty acids (SFA) and diets with a high glycemic index (GI) have been shown to increase liver fat content. However, available data from human dietary intervention studies is limited and these studies did not reflect a realistic diet. Here the investigators want to combine low GI/SFA on the one hand and high GI/SFA on the other hand to reflect realistically a healthy and an unhealthy diet as they are actually consumed by the Dutch population. It is hypothesized that such a low compared to a high GI/SFA diet reduces liver fat content and possibly liver fat composition. Furthermore, underlying pathways involved in mediating those changes in liver fat are largely unknown. Hepatic lipid storage can originate from several metabolic pathways, including de novo lipogenesis (DNL) or decreased hepatic fat oxidation. Based on current literature the investigators hypothesize that with the diets chosen here, both DNL (by differences in GI) and fat oxidation (by differences in fat composition) will be involved in causing changes in liver fat.

Objective:

The primary objective of this study is to investigate whether a two-week low compared to high GI/SFA diet reduces liver fat content. In addition, it will be investigated whether a two- week low compared to high GI/SFA diet reduces DNL, lowers the 24-hour glycemic response, lowers hepatic glycogen content, increases hepatic fat oxidation and changes hepatic lipid composition. Furthermore, the metabolic response to a meal (metabolites related to energy metabolism and substrate oxidation) will be studied upon the low and high GI/SFA diets.

Study design:

This is a randomized cross-over study comparing the effects of a high GI/SFA compared to a low GI/SFA diet.

Study population:

Up to seventeen healthy overweight/obese males and postmenopausal females, aged between 45-75 years and BMI between 27-38 kg/m2 will participate in the study (minimally 13 volunteers need to finish the study).

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* Male or postmenopausal female
* Aged 45-75 years at start of the study
* Body mass index (BMI) 27 - 38 kg/m2
* Stable dietary habits (no weight loss or gain >3kg in the past 3 months) Sedentary lifestyle (not more than 2 hours of sports per week)
* TG between 1.0 and 4.0 mmol/L

Exclusion Criteria:

* Type 2 diabetes
* Any acute condition, exacerbation of chronic condition, or medical history that would in the investigator's or dependent physician's opinion interfere with the study
* Contra-indication for MRI (which can be found in appendix II)
* Alcohol consumption of >2 servings per day
* Smoking
* Use of medication known to interfere with the safety of study procedures

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-03-23 (Actual)

PRIMARY OUTCOMES:
Hepatic fat content | 20 minutes
  Expressed as a percentage, measured by 1H-MRS

SECONDARY OUTCOMES:
Hepatic De Novo Lipogenesis | 20 hours
  Percentage of palmitate in VLDL-TG originating from DNL
Hepatic fat composition (%SFA, MUFA, PUFA) | 20 minutes
  Measured by 1H-MRS
Hepatic glycogen content | 20 minutes
  Measured by 13C-MRS

CONTACTS AND LOCATIONS:
Overall Officials: Vera Schrauwen-Hinderling, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No